CLINICAL TRIAL: NCT03194776
Title: A Patient and Investigator-blinded, Randomized, Placebo Controlled Study of LLG783 in Patients With Peripheral Artery Disease (PAD) and Intermittent Claudication
Brief Title: Study of LLG783 in Patients With Peripheral Artery Disease (PAD) and Intermittent Claudication
Acronym: PAD PoC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CLLG783X2201; 2017-000706-37 (EudraCT Number)
Record Dates: First submitted 2017-06-19; First posted 2017-06-21 (Actual); Results first posted 2020-01-31 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2020-03

CONDITIONS: Peripheral Artery Disease (PAD); Intermittent Claudication
Keywords: PAD; peripheral artery/arterial disease; peripheral vascular disease; leg pain; claudication; leg pain with exercise; exercise test; walk test
MeSH Terms: conditions — Peripheral Arterial Disease; Intermittent Claudication; Peripheral Vascular Diseases

STUDY DESIGN:
Intervention Model Description: Randomized, patient and investigator-blinded, placebo controlled, parallel group study
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- LLG783 (Experimental): Patients will receive LLG783 i.v. infusion every 4 weeks for 12 weeks.
  Interventions: Drug: LLG783
- Placebo (Placebo Comparator): Patients will receive placebo to LLG783 i.v. infusion every 4 weeks for 12 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LLG783 — LLG783 concentrate solution for infusion/injection suitable for i.v. administration as well as s.c. administration.
  Arms: LLG783
Drug: Placebo — Placebo to LLG783 concentrate solution for infusion/injection suitable for i.v. administration as well as s.c. administration.
  Arms: Placebo

SUMMARY:
This study is designed to determine whether LLG783 displays the clinical safety and efficacy profile, after multiple i.v. doses, to support further development in patients with PAD and intermittent claudication.

ELIGIBILITY:
Inclusion Criteria:

* claudication, as defined by pain with exertion in either leg;
* On stable medical therapy, including statins, aspirin, and antihypertensive medications (as medically indicated) unless individually contraindicated, for at least 4 weeks prior to the screening visit;
* Vital signs must be within the following ranges:

  * body temperature between 35.0-37.5°C
  * systolic blood pressure, 90-159 mm Hg
  * diastolic blood pressure, 50-99 mm Hg
  * pulse rate, 50 - 90 bpm
* Moderately impaired ambulatory function judged by the investigator to be due primarily to PAD and assessed by a maximum walk distance between 50 and 400 meters (inclusive of these values) at the screening 6-minute walk test (6MWT).

Exclusion Criteria:

* Pregnant or nursing (lactating) women;
* Patients who meet any of the following PAD related criteria:

  * Patients actively attending and participating in a supervised exercise rehabilitation program (patients who have already completed such a program and remain symptomatic may be included).
  * Patients with any condition other than PAD that limits walking ability.
  * Known inflammatory disease of the arteries (other than atherosclerosis; e.g. Thromboangiitis obliterans).
  * Clinical evidence of critical limb ischemia including new or non-healing ulcers (felt secondary to critical limb ischemia), new or recent onset of resting pain in the lower extremities particularly at night (felt secondary to critical limb ischemia) and/or gangrene of the lower extremities (Fontaine stage III-IV) .
* Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using highly effective methods of contraception during dosing and for 150 days after stopping of investigational drug.
* Any of the following concomitant cardiovascular or metabolic conditions or diseases:

  * Myocardial infarction within 6 months of screening.
  * Stroke within 6 months of screening.
  * History of clinically significant ventricular arrhythmias, according to the discretion of the investigator, within 6 months of screening.
  * Significant ECG abnormalities, according to the discretion of the investigator, at screening.
  * History of sustained and clinically significant supraventricular arrhythmias (e. g. associated with hemodynamic compromise) within 6 months of screening.
  * Chronic heart failure New York Heart Association Class III or IV.
  * Known presence of aortic aneurysm > 5 cm.
  * Uncontrolled diabetes as defined by a random fasting glucose level of 13 mmol/L or 240 mg/dL or a HbA1c greater than 9% as measured at screening. Diabetes should be treated as appropriate during the study.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2017-09-20 (Actual); Primary Completion 2018-09-07 (Actual); Study Completion 2018-12-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (6):
- United States (2):
  - Novartis Investigative Site, Jacksonville, Florida
  - Novartis Investigative Site, Columbus, Ohio
- Germany (3):
  - Novartis Investigative Site, Kiel, Schleswig-Holstein
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Magdeburg
- Novartis Investigative Site, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- See also: A Plain Language Trial Summary is available on novartisclinicatrials.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=474

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 46 subjects with clinical evidence of PAD and intermittent claudication were enrolled and randomized in this study.
Groups:
- LLG783 6mg/kg: Participants received LLG783 6 milligram per kilogram (mg/kg) as intravenous (IV) infusion once every 4 weeks for a total of 4 doses over a period of 12 weeks.
- Placebo: Participants received placebo as IV infusion once every 4 weeks for a total of 4 doses over a period of 12 weeks.
Period: Overall Study
Arm/Group | LLG783 6mg/kg | Placebo
Started | 23 | 23
Completed | 23 | 23
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- LLG783 6mg/kg: Participants received LLG783 6 mg/kg as IV infusion once every 4 weeks for a total of 4 doses over a period of 12 weeks.
- Total: Total of all reporting groups
Arm/Group | LLG783 6mg/kg | Placebo | Total
Number analyzed (Participants) | 23 | 23 | 46
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.0 (7.1) | 66.3 (6.9) | 66.7 (6.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 5 | 13
  Male | 15 | 18 | 33
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 23 | 23 | 46
  Unknown or Not Reported | 0 | 0 | 0
Maximum walking distance (MWD) [Mean (Standard Deviation); unit: meters] — MWD was determined by 6-minute walking test (6-MWT), an exercise test measuring the distance walked by a participant over a span of 6 minutes.
  meters | 317.3 (62.0) | 311.3 (84.0) | 314.3 (73.0)
Pain Free Walking Distance (PWFD) [Mean (Standard Deviation); unit: meters] — PWFD was defined as the distance walked up to the point of onset of claudication symptoms (pain) recorded during the 6MWT.
  meters | 160.7 (79.4) | 156.0 (86.7) | 158.3 (82.3)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs), Drug-related AEs, Serious Adverse Events (SAEs) and Deaths
Description: An AE is any untoward medical occurrence (that is, any unfavorable and unintended sign, including abnormal laboratory findings, symptom or disease) in a participant after providing written informed consent for participation in the study until the end of study visit. Therefore, an AE may or may not be temporally or causally associated with the use of a medicinal (investigational) product. An SAE is defined as any AE which is is fatal or life-threatening, results in persistent or significant disability/incapacity, constitutes a congenital anomaly/birth defect in offspring, requires inpatient hospitalization or prolongation of existing hospitalization and is is medically significant.
Time Frame: Up to 32 Weeks
Population: Safety analysis set included all participants that received any study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | LLG783 6mg/kg | Placebo
Number analyzed (Participants) | 23 | 23
Participants
  AEs | 18 | 17
  Drug-related AEs | 4 | 4
  SAEs | 1 | 2
  Death | 0 | 0

2. Primary Outcome: Change From Baseline in Maximum Walking Distance (MWD) as Assessed by 6-minute Walk Test (6MWT) at Week 16
Description: MWD was assessed by the 6MWT prior to dosing was used to evaluate functional capacity of peripheral artery disease (PAD) participants. 6MWT test included measurement of total distance walked in 6 minutes.
Time Frame: Baseline, Week 16 (Day 113)
Population: Pharmacodynamic (PD) analysis set included all participants with available PD data, who received any study treatment and experienced no protocol deviations with relevant impact on PD data. Here 'N' (overall number of participants analyzed) signifies number of participants evaluable for this endpoint.
Measure: Least Squares Mean (80% Confidence Interval); unit: meter (m)
Arm/Group | LLG783 6mg/kg | Placebo
Number analyzed (Participants) | 22 | 19
meter (m) | 19.10 [5.30 to 32.90] | 36.84 [21.99 to 51.70]
Statistical Analysis 1: Comparison: LLG783 6mg/kg vs Placebo; Statistical analysis was done by mixed effect model repeat measurement (MMRM) model analysis; Test type: Superiority; p = 0.2612, two-sided test — P-value of <= 0.2 was considered significant; Mean Difference (Final Values) = -17.74, 80% CI 2-sided [-38.03 to 2.55]

3. Secondary Outcome: Area Under the Serum Concentration-time Curve From Time Zero to Infinity (AUCinf)
Description: AUCinf is defined as the area under the serum concentration-time curve from time zero to infinity.
Time Frame: 1 hour predose and 1, 2 and 4 hours postdose on Day 1; 0 hour predose and 1, 2 and 4 hours postdose on Day 85
Population: PK analysis set: Participants with at least 1 available valid PK concentration measurement, who received any study treatment and with no protocol deviations that impacted PK data. N (overall number of participants analyzed) = participants evaluable for this outcome measure and 'n' (number analyzed) = participants evaluable at specified time points.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: day*microgram per millileter (day*mg/mL)
Groups:
- LLG783 6 mg/kg: Participants received LLG783 6 mg/kg as IV infusion once every 4 weeks for a total of 4 doses over a period of 12 weeks.
Arm/Group | LLG783 6 mg/kg
Number analyzed (Participants) | 20
day*microgram per millileter (day*mg/mL)
  Day 1 | 2110 (21.1)
  Day 85 | 4860 (39.1)

4. Secondary Outcome: Area Under the Serum Concentration-time Curve From Time Zero to the Time of the Last Quantifiable Concentration (AUClast)
Description: AUClast is defined as the area under the serum concentration-time curve from time zero to the time of the last quantifiable concentration.
Time Frame: 1 hour predose and 1, 2 and 4 hours postdose on Day 1; 0 hour predose on Day 29 and 57; 0 hour predose and 1, 2 and 4 hours postdose on Day 85
Population: Pharmacokinetic (PK) analysis set included all participants with at least one available valid PK concentration measurement, who received any study treatment and with no protocol deviations that impacted PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: day*mcg/mL
Arm/Group | LLG783 6 mg/kg
Number analyzed (Participants) | 23
day*mcg/mL
  Day 1 | 1660 (33.6)
  Day 85 | 4930 (38.9)

5. Secondary Outcome: Area Under the Serum Concentration-time Curve From Time Zero to Defined Time Point 't' (AUC[0-t])
Description: AUC(0-t)is defined as the area under the serum concentration-time curve from time zero to time 't' where is a defined time point after administration.
Time Frame: as for outcome 4
Population: PK analysis set included all participants with at least one available valid PK concentration measurement, who received any study treatment and with no protocol deviations that impacted PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: day*mcg/mL
Arm/Group | LLG783 6 mg/kg
Number analyzed (Participants) | 23
day*mcg/mL
  Day 1 | 1640 (34.1)
  Day 85 | 3130 (34.7)

6. Secondary Outcome: Area Under the Serum Concentration-time Curve From Time Zero to the End of the Dosing Interval Tau (AUCtau)
Description: AUCtau is defined as the area under the serum concentration-time curve from time zero to the end of the dosing interval tau.
Time Frame: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: day*mcg/mL
Arm/Group | LLG783 6 mg/kg
Number analyzed (Participants) | 23
day*mcg/mL
  Day 1 | 1640 (34.1)
  Day 85 | 3130 (34.7)

7. Secondary Outcome: Observed Maximum Serum Concentration (Cmax) Following Drug Administration
Description: Cmax is defined as the observed maximum serum concentration following drug administration.
Time Frame: as for outcome 4
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram per milliliter (mcg/mL)
Arm/Group | LLG783 6 mg/kg
Number analyzed (Participants) | 23
microgram per milliliter (mcg/mL)
  Day 1 | 203 (40.0)
  Day 85 | 268 (39.8)

8. Secondary Outcome: Time to Reach the Maximum Concentration After Drug Administration (Tmax)
Description: Tmax is defined as the time to reach the maximum concentration after drug administration.
Time Frame: as for outcome 4
Population: as for outcome 5
Measure: Median (Full Range); unit: Days
Arm/Group | LLG783 6 mg/kg
Number analyzed (Participants) | 23
Days
  Day 1 | 0.0833 [0.0417 to 3.01]
  Day 85 | 0.0833 [0.0431 to 9.94]

9. Secondary Outcome: Change From Baseline in Pain-free Walking Distance (PFWD) as Assessed by 6-minute Walk Test at Week 16
Description: PFWD was defined as the distance walked up to the point of onset of claudication symptoms (pain) recorded during the 6MWT and was used to evaluate symptomatic functional capacity of PAD participants. The PFWD was measured as the distance walked up to the time/place where the participant first experiences symptoms typical of their claudication which included pain, cramps, or other discomfort in the buttocks, thighs, calves or feet that occurs during the 6MWT exercise period.
Time Frame: Baseline, Week 16 (Day 113)
Population: PD analysis set included all participants with available PD data, who received any study treatment and experienced no protocol deviations with relevant impact on PD data. Here 'N' (overall number of participants analyzed) signifies number of participants evaluable for this outcome measure.
Measure: Least Squares Mean (80% Confidence Interval); unit: meters
Arm/Group | LLG783 6mg/kg | Placebo
Number analyzed (Participants) | 22 | 19
meters | 44.77 [20.52 to 69.02] | 57.09 [30.97 to 83.22]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from first dose of study treatment until end of study treatment, plus 30 days post treatment, up to maximum duration of approximately 15 months.
Description: Any sign or symptom that occurs during the study treatment plus the 30 days post treatment.
Groups:
- LLG783 i.v. 6 mg/kg: Participants received LLG783 6 mg/kg as IV infusion once every 4 weeks for a total of 4 doses over a period of 12 weeks.
Arm/Group | LLG783 i.v. 6 mg/kg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/23
Serious Adverse Events (participants affected / at risk) | 1/23 | 2/23
Other Adverse Events (participants affected / at risk) | 18/23 | 16/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LLG783 i.v. 6 mg/kg (N=23) | Placebo (N=23)
Hypochromic anaemia (Blood and lymphatic system disorders) | 1 | 0
Gastritis haemorrhagic (Gastrointestinal disorders) | 0 | 1
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LLG783 i.v. 6 mg/kg (N=23) | Placebo (N=23)
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Hypochromic anaemia (Blood and lymphatic system disorders) | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1
Atrial flutter (Cardiac disorders) | 1 | 0
Bradycardia (Cardiac disorders) | 0 | 2
Pericardial effusion (Cardiac disorders) | 1 | 0
Sinus bradycardia (Cardiac disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 3 | 1
Nausea (Gastrointestinal disorders) | 1 | 0
Toothache (Gastrointestinal disorders) | 1 | 0
Fatigue (General disorders) | 2 | 1
Medical device site irritation (General disorders) | 3 | 0
Oedema peripheral (General disorders) | 2 | 0
Peripheral swelling (General disorders) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0
Cystitis (Infections and infestations) | 1 | 0
Erysipelas (Infections and infestations) | 0 | 1
Infected bite (Infections and infestations) | 0 | 1
Nasopharyngitis (Infections and infestations) | 5 | 4
Paronychia (Infections and infestations) | 1 | 0
Root canal infection (Infections and infestations) | 0 | 1
Tooth abscess (Infections and infestations) | 1 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 1 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Thermal burn (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0
Blood creatinine increased (Investigations) | 1 | 0
Blood pressure increased (Investigations) | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 0
Weight increased (Investigations) | 1 | 0
Iron deficiency (Metabolism and nutrition disorders) | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Carpal tunnel syndrome (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 2 | 2
Neuralgia (Nervous system disorders) | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 2
Sciatica (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Adjustment disorder with depressed mood (Psychiatric disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1
Stasis dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 1
Peripheral arterial occlusive disease (Vascular disorders) | 3 | 1
Peripheral ischaemia (Vascular disorders) | 0 | 1
Spider vein (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of pooled data (i.e.,data from all sites) in clinical trial or disclosure of trial results in their entirety.

DOCUMENTS (2):
  • Study Protocol (2017-11-01): https://cdn.clinicaltrials.gov/large-docs/76/NCT03194776/Prot_000.pdf
  • Statistical Analysis Plan (2019-02-08): https://cdn.clinicaltrials.gov/large-docs/76/NCT03194776/SAP_001.pdf